CLINICAL TRIAL: NCT02065401
Title: A Phase 1, Open-label, Randomized, 3-Period, Relative Bioavailability Study Comparing the Pharmacokinetics of Granule and Tablet Formulations of Deferitazole (Disodium Salt) and a Capsule Formulation of Deferitazole (Magnesium Hydroxide Salt), Each Administered as a Single Oral Dose
Brief Title: Pharmacokinetics of Granule and Tablet Formulations of Deferitazole (Disodium Salt) and a Capsule Formulation of Deferitazole (Magnesium Hydroxide Salt)
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: This study was withdrawn until the evaluation of the nonclinical rat findings is complete.
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: SPD602-112
Record Dates: First submitted 2014-02-10; First posted 2014-02-19 (Estimated); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Healthy
MeSH Terms: interventions — Tablets

ARMS (3):
- Deferitazole (disodium salt, granule) (Experimental)
  Interventions: Drug: Deferitazole (disodium salt, granule)
- Deferitazole (disodium salt, tablet) (Experimental)
  Interventions: Drug: Deferitazole (disodium salt, tablet)
- Deferitazole (magnesium hydroxide salt) (Experimental)
  Interventions: Drug: Deferitazole (magnesium hydroxide salt)

INTERVENTIONS:
Drug: Deferitazole (disodium salt, granule) — Single oral dose of 1500 mg administered on Day 1
  Other Names: SPD602, SSP-004184, SSP-004184SS
  Arms: Deferitazole (disodium salt, granule)
Drug: Deferitazole (disodium salt, tablet) — Single oral dose of 1500 mg administered on Day 1
  Other Names: SPD602, SSP-004184, SSP-004184SS
  Arms: Deferitazole (disodium salt, tablet)
Drug: Deferitazole (magnesium hydroxide salt) — Single oral dose of 2400 mg administered on Day 1
  Other Names: SPD602, SSP-004184AQ, SSP-004184
  Arms: Deferitazole (magnesium hydroxide salt)

SUMMARY:
The purpose of this study is to compare the pharmacokinetic profiles of deferitazole after administration of granule and tablet formulations of a deferitazole disodium salt to a capsule formulation of deferitazole magnesium hydroxide salt (reference formulation) in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years inclusive at the time of consent.
2. Must be considered "healthy".
3. Serum ferritin, hemoglobin and erythrocyte indices (packed cell volume, mean corpuscular volume and mean corpuscular hemoglobin concentration) within normal range.
4. Willingness to comply with any applicable contraceptive requirements of the protocol and is:

   * Male, or
   * Female of non-childbearing potential (defined as a female who is post-menopausal )
   * Non-pregnant, non-lactating female
   * Females must be at least 90 days post partum or nulliparous.
5. Body weight equal to or greater than 60kg.
6. Ability to swallow a dose of the investigational product.

Exclusion Criteria:

1. Subject has a clinically significant history or a disorder detected during the medical interview/physical examination.
2. Acute illness.
3. Oral condition:

   * Has history of oral surgery (including extractions) within 4 weeks, operative dental work within 7 days, or a presence of any clinically significant oral pathology (as determined by the investigator) including lesions, sores or inflammation which would interfere with assessments.
   * Has fixed retainers, orthodontic appliances, or either maxillary and/or mandibular dentures or other appliances which may interfere with swilling or tasting the formulations.
   * Has current or recurrent disease that could affect the mouth and interfere with the taste assessment.
   * Has severe gingivitis, periodontitis or rampant caries.
   * Has the presence of oral or peri-oral ulceration including herpetic lesions
   * Has elective dentistry scheduled during the study duration.
4. Subject has a history of thyroid disorder that has not been stabilized on thyroid medication or treatment.
5. History of alcohol or other substance abuse within the year.
6. A positive screen for alcohol or drugs of abuse.
7. Confirmed systolic blood pressure >139mmHg or <89mmHg, and diastolic blood pressure >89mmHg or<49mmHg.
8. Routine consumption of more than 2 units of caffeine per day or subjects who experience caffeine withdrawal headaches.
9. Male subjects who consume more than 3 units of alcohol per day. Female subjects who consume more than 2 units of alcohol per day.
10. A positive human immunodeficiency virus antibody screen, hepatitis B surface antigen, or hepatitis C virus antibody.
11. Current use of any other medication (including over-the-counter, herbal, or homeopathic preparations)
12. Current use of iron supplements and/or multivitamins.
13. Use of tobacco in any form (e.g., smoking or chewing) or other nicotine-containing products.
14. Donation of blood or blood products (e.g., plasma or platelets) within 60 days.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-02-28 (Estimated); Primary Completion 2014-03-19 (Estimated); Study Completion 2014-03-19 (Estimated)

PRIMARY OUTCOMES:
Area Under the Plasma Concentration-time Curve (AUC) of Deferitazole | Up to 120 hours post-dose
  AUC of disodium salt granule, disodium salt tablet, and magnesium hydroxide salt
Maximum Plasma Concentration (Cmax) of Deferitazole | Up to 120 hours post-dose
  Cmax of disodium salt granule, disodium salt tablet, and magnesium hydroxide salt

SECONDARY OUTCOMES:
Taste of Deferitazole | Immediately after dose and 5 minutes post-dose
Bioequivalence of Deferitazole Disodium Salt Granule Formulation With Tablet Formulation | Up to 120 hours post-dose
  Compare the pharmacokinetic profile of granule formulation with pharmacokinetic profile of tablet formulation

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Clinical Pharmacology of Miami, Miami, Florida, United States